CLINICAL TRIAL: NCT01923389
Title: A Phase 1, Placebo-Controlled, Randomized Trial To Assess The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Multiple Intravenous Doses Of PF-05231023 In Obese Adult Subjects
Brief Title: Multiple Dose Study Of PF-05231023 In Obese Adult Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated on December 19th, 2013 due to a business decision by the Sponsor. No safety concerns have been observed in this study.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: B2901009
Record Dates: First submitted 2013-07-30; First posted 2013-08-15 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: T2DM; obesity; safety; multiple dose; intravenous
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — PF-05231023

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- 100 mg PF-05231023 (Experimental)
  Interventions: Drug: 100 mg PF-05231023

INTERVENTIONS:
Other: Placebo — 0.9% w/v sodium chloride injection, United States Pharmacopeia (USP), twice a week for 4 weeks.
  Arms: Placebo
Drug: 100 mg PF-05231023 — 100 mg IV infusion twice a week for 4 weeks
  Arms: 100 mg PF-05231023

SUMMARY:
This is a trial in obese subjects to study the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple doses of PF-05231023.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects of non-childbearing potential between the ages of 21 and 70.
* Subjects with a BMI of 30 to 45.4 kg/m2 and total body weight >110 lbs.

Exclusion Criteria:

* Recent (6 months) unstable concurrent disease.
* History of allergic disease or drug allergies.
* Any condition affecting food consumption or absorption.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Orlando, Florida, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2901009&StudyName=Multiple%20Dose%20Study%20Of%20PF-05231023%20In%20Obese%20Adult%20Subjects

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo (normal saline) was administered as a 20-milliliters (mL) intravenous (IV) infusion twice weekly on Days 1, 4, 8, 11, 15, 18, 22 and 25.
- PF-05231023 100 mg: PF-05231023 100 mg was administered as a 20-mL IV infusion twice weekly on Days 1, 4, 8, 11, 15, 18, 22 and 25.
Period: Overall Study
Arm/Group | Placebo | PF-05231023 100 mg
Started | 2 | 2
Completed | 1 | 2
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study medication (PF-05231023 or placebo).
Groups:
- Placebo: Placebo (normal saline) was administered as a 20-mL IV infusion twice weekly on Days 1, 4, 8, 11, 15, 18, 22 and 25.
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-05231023 100 mg | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (4.2) | 34.0 (5.7) | 36.5 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AEs were also reported for the 7-day pre-randomization period.
Time Frame: Day -7 through the last follow-up (Day 68)
Population: All participants who received at least 1 dose of study medication (PF-05231023 or placebo).
Measure: Number; unit: Participants
Arm/Group | Placebo | PF-05231023 100 mg
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

2. Primary Outcome: Number of Participants With Vital Signs Data Met Criteria of Potential Clinical Concern
Description: Vital signs included supine systolic blood pressure, diastolic blood pressure and pulse rate. Vital signs criteria of potential clinical concern were 1), blood pressure: systolic greater than or equal to (>=)30 millimeters of mercury (mm Hg) change from baseline in the same posture or systolic less than (<)90 mm Hg; diastolic >=20 mm Hg change from baseline in the same posture or diastolic <50 mm Hg; 2), Pulse rate: supine/Sitting: <40 or greater than (>) 120 beats per minute (bpm); Standing: <40 or >140 bpm.
Time Frame: Days -7 up to the last follow-up (Day 68)
Population: All participants who received at least 1 dose of study medication (PF-05231023 or placebo).
Measure: Number; unit: Participants
Arm/Group | Placebo | PF-05231023 100 mg
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Data Met Criteria of Potential Clinical Concern
Description: ECG criteria of potential clinical concern were 1), PR interval:>=300 msec, >=25% increase when baseline >200 msec, or >=50% increase when baseline <=200 msec; 2), QRS interval:>=140 msec, or >=50% increase from baseline; 3), QT interval corrected for heart rate (QTc)/QTc interval using Fridericia's formula (QTcF):>=500 msec, QTcF interval: absolute value >=450 - <480 msec(borderline), >=480 msec (prolonged), absolute change 30 - <60 msec (borderline) or >=60 msec (prolonged). 12-lead ECG (triplicate) was performed on Day 0 and 12-lead ECG (singlet) was performed at other times.
Time Frame: Days -7 up to the last follow-up (Day 68)
Population: All participants who received at least 1 dose of study medication (PF-05231023 or placebo).
Measure: Number; unit: Participants
Arm/Group | Placebo | PF-05231023 100 mg
Number analyzed (Participants) | 2 | 2
Participants | 1 | 0

4. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Measurements
Description: The total number of participants with laboratory test abnormalities without regard to baseline abnormality was assessed.
Time Frame: Days -7 up to the last follow-up (Day 68)
Population: All participants who received at least 1 dose of study medication (PF-05231023 or placebo).
Measure: Number; unit: Participants
Arm/Group | Placebo | PF-05231023 100 mg
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

5. Primary Outcome: Number of Participants With Positive Anti-PF-05231023 Antibodies and Neutralizing Antibodies.
Description: Anti-PF-05231023 antibodies were analyzed using a tiered testing strategy of screen, confirm, and titer characterization. Positive was defined as titer value >=6.23 and negative was defined as titer value <6.23. Samples tested positive were also to be analyzed in a neutralization assay to determine whether or not they were neutralizing or non-neutralizing.
Time Frame: Days 1 up to the last follow-up (Day 68)
Population: All participants who received at least 1 dose of active study medication (PF-05231023). Neutralizing antibodies were not tested because all participants who received PF-05231023 100 mg tested negative for anti-PF-05231023 antibodies.
Measure: Number; unit: Participants
Arm/Group | Placebo | PF-05231023 100 mg
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

6. Secondary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Tau, the Dosing Interval (AUCtau) of PF-05231023 (C-terminus and N-terminus PF-05231023 and Total CVX-2000 Antibody Scaffold)
Time Frame: Days 1 and 25
Population: AUCtau for C-terminus and N-terminus of PF-05231023 and CVX-2000 were not summarized due to the premature termination of the study.
Arm/Group | PF-05231023 100 mg
Number analyzed (Participants) | 0

7. Secondary Outcome: Maximum Plasma Concentration (Cmax) of PF-05231023 (C-terminus and N-terminus PF-05231023 and Total CVX-2000 Antibody Scaffold)
Time Frame: Days 1 and 25
Population: Cmax for C-terminus and N-terminus of PF-05231023 and CVX-2000 were not summarized due to the premature termination of the study.
Arm/Group | PF-05231023 100 mg
Number analyzed (Participants) | 0

8. Secondary Outcome: Lowest Concentration Observed During Dosing Interval (Cmin) of PF-05231023 (C-terminus and N-terminus PF-05231023 and Total CVX-2000 Antibody Scaffold)
Time Frame: Day 25
Population: Cmin for C-terminus and N-terminus of PF-05231023 and CVX-2000 were not summarized due to the premature termination of the study.
Arm/Group | PF-05231023 100 mg
Number analyzed (Participants) | 0

9. Secondary Outcome: Average Concentration at Steady State (Cav) of PF-05231023 (C-terminus and N-terminus PF-05231023 and Total CVX-2000 Antibody Scaffold)
Time Frame: Day 25
Population: Cav for C-terminus and N-terminus of PF-05231023 and CVX-2000 were not reported due to the premature termination of the study.
Arm/Group | PF-05231023 100 mg
Number analyzed (Participants) | 0

10. Secondary Outcome: Time for Cmax (Tmax)of PF-05231023 (C-terminus and N-terminus PF-05231023 and Total CVX-2000 Antibody Scaffold)
Time Frame: Day 25
Population: Tmax for C-terminus and N-terminus of PF-05231023 and CVX-2000 were not summarzied due to the premature termination of the study.
Arm/Group | PF-05231023 100 mg
Number analyzed (Participants) | 0

11. Secondary Outcome: Clearance (CL)of PF-05231023 (C-terminus and N-terminus PF-05231023 and Total CVX-2000 Antibody Scaffold)
Time Frame: Day 25
Population: CL for C-terminus and N-terminus of PF-05231023 and CVX-2000 were not summarzied due to the premature termination of the study.
Arm/Group | PF-05231023 100 mg
Number analyzed (Participants) | 0

12. Secondary Outcome: Terminal Elimination Half-life (t1/2)of PF-05231023 (C-terminus and N-terminus PF-05231023 and Total CVX-2000 Antibody Scaffold)
Time Frame: Day 25
Population: t1/2 for C-terminus and N-terminus of PF-05231023 and CVX-2000 were not summarzied due to the premature termination of the study.
Arm/Group | PF-05231023 100 mg
Number analyzed (Participants) | 0

13. Secondary Outcome: Observed Accumulation Ratio (Rac) for Cmax and AUCtau of PF-05231023 (C-terminus and N-terminus PF-05231023 and Total CVX-2000 Antibody Scaffold)
Time Frame: Day 25
Population: Rac for C-terminus and N-terminus of PF-05231023 and CVX-2000 were not summarzied due to the premature termination of the study.
Arm/Group | PF-05231023 100 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Day -7 through Day 68 (AEs occurred after first dose of study drug were treatment-emergent). Serious AEs (SAEs) were reported from time that subject provided informed consent until 28 calendar days after last dose of the study drug.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | PF-05231023 100 mg
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2) | PF-05231023 100 mg (N=2)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 — Treatment-emergent
Diarrhoea (Gastrointestinal disorders) | 0 | 1 — Treatment-emergent
Eructation (Gastrointestinal disorders) | 0 | 1 — Treatment-emergent
Flatulence (Gastrointestinal disorders) | 1 | 0 — Treatment-emergent
Nausea (Gastrointestinal disorders) | 0 | 1 — Treatment-emergent
Chest pain (General disorders) | 1 | 0 — Treatment-emergent
Chills (General disorders) | 0 | 1 — Treatment-emergent
Puncture site pain (General disorders) | 1 | 0 — Treatment-emergent
Upper respiratory tract infection (Infections and infestations) | 1 | 0 — Treatment-emergent
Laceration (Injury, poisoning and procedural complications) | 0 | 1 — Treatment-emergent
Wound (Injury, poisoning and procedural complications) | 0 | 1 — Treatment-emergent
Headache (Nervous system disorders) | 1 | 0 — Treatment-emergent
Hypoaesthesia (Nervous system disorders) | 0 | 1 — Treatment-emergent
Middle insomnia (Psychiatric disorders) | 1 | 0 — Treatment-emergent
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Treatment-emergent
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Treatment-emergent
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Treatment-emergent
Contusion (Injury, poisoning and procedural complications) | 0 | 1 — Events during pre-randomization 7-day diet run-in period
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 — Events during pre-randomization 7-day diet run-in period
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Events during pre-randomization 7-day diet run-in period

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.